CLINICAL TRIAL: NCT03290196
Title: The Effect of EXPAREL® on Postsurgical Pain, and the Use of Narcotics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients pain was not regulated well with this product.
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXPAREL
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tear
Keywords: Shoulder; Rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXPAREL 1.3 % in 20 ML Injection (Other): EXPAREL (bupivacaine liposome injectable suspension, 20 mL single use vial, 1.3% [13.3 mg/mL]) is a liposome injection of bupivacaine, an amide local anesthetic, indicated for single-dose infiltration into the surgical site to produce postsurgical analgesia. EXPAREL dosage is based on the following factors:
  * size of surgical site
  * volume required to cover the area
  * individual patient factors that may impact the safety of an amide local anesthetic
  * maximum doe of 266 mg (20 mL)
  Interventions: Drug: EXPAREL 1.3 % in 20 ML Injection

INTERVENTIONS:
Drug: EXPAREL 1.3 % in 20 ML Injection — EXPAREL single shot dose given as an analgesia for arthroscopic rotator cuff repair surgery.
  Other Names: bupivacaine liposome injectable suspension

SUMMARY:
Patients undergoing shoulder rotator cuff surgery in an outpatient setting are the focus of this study. The purpose of this study is to determine if the product EXPAREL® can be used as a safe alternative in shoulder surgery to pain pumps, while limiting narcotic use and providing appropriate postoperative pain control.

DETAILED DESCRIPTION:
Based on prior research, it is hypothesized EXPAREL® can potentially be used as a local anesthetic option after undergoing an arthroscopic rotator cuff repair in the outpatient setting. Conducting this study, will allow the option for a surgeon to administer a local anesthetic, in a single injection, to the exact location of the surgical procedure and in a sterile environment. The purpose of this pilot study is to determine if EXPAREL® can be used as a safe alternative to current post-operative pain control methods, while limiting narcotic use and providing appropriate postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-72 years of age
* Subjects scheduled to undergo a rotator cuff repair with a subacromial decompression by one of the protocol investigators

Exclusion Criteria:

* Planned concomitant glenoid labral repair
* Previous open shoulder surgery
* Neurological deficit or other disability involving the surgical extremity
* Anyone with a documented allergy to bupivicaine
* Subjects that are not mentally competent to give consent
* Pregnant women
* Subjects with an intolerance to hydrocodone or oxycodone and/or brand name equivalent combination medication

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Andrews, MD, Principal Investigator — Andrews Institute for Orthopaedics & Sports Medicine
Locations (1):
- Andrews Research & Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson MD, Mickler T, Arthur GR, Rosenburg S, Wilson R. Bupivacaine with and without epinephrine for intercostal nerve block. J Cardiothorac Anesth. 1990 Apr;4(2):200-3. doi: 10.1016/0888-6296(90)90238-b. PMID 2131867
- [Background] Colombo G, Padera R, Langer R, Kohane DS. Prolonged duration local anesthesia with lipid-protein-sugar particles containing bupivacaine and dexamethasone. J Biomed Mater Res A. 2005 Nov 1;75(2):458-64. doi: 10.1002/jbm.a.30443. PMID 16088895
- [Background] Bergese SD, Onel E, Morren M, Morganroth J. Bupivacaine extended-release liposome injection exhibits a favorable cardiac safety profile. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):145-51. doi: 10.1097/AAP.0b013e31823d0a80. PMID 22266897
- [Background] Portillo J, Kamar N, Melibary S, Quevedo E, Bergese S. Safety of liposome extended-release bupivacaine for postoperative pain control. Front Pharmacol. 2014 Apr 30;5:90. doi: 10.3389/fphar.2014.00090. eCollection 2014. PMID 24817851
- [Background] Candiotti K. Liposomal bupivacaine: an innovative nonopioid local analgesic for the management of postsurgical pain. Pharmacotherapy. 2012 Sep;32(9 Suppl):19S-26S. doi: 10.1002/j.1875-9114.2012.01183.x. PMID 22956491
- [Background] Cohen SM, Vogel JD, Marcet JE, Candiotti KA. Liposome bupivacaine for improvement in economic outcomes and opioid burden in GI surgery: IMPROVE Study pooled analysis. J Pain Res. 2014 Jun 24;7:359-66. doi: 10.2147/JPR.S63764. eCollection 2014. PMID 25018650
- [Background] Bagsby DT, Ireland PH, Meneghini RM. Liposomal bupivacaine versus traditional periarticular injection for pain control after total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1687-90. doi: 10.1016/j.arth.2014.03.034. Epub 2014 Apr 4. PMID 24793570
- [Background] Singelyn FJ, Lhotel L, Fabre B. Pain relief after arthroscopic shoulder surgery: a comparison of intraarticular analgesia, suprascapular nerve block, and interscalene brachial plexus block. Anesth Analg. 2004 Aug;99(2):589-92, table of contents. doi: 10.1213/01.ANE.0000125112.83117.49. PMID 15271745
- [Background] Borgeat A, Ekatodramis G, Kalberer F, Benz C. Acute and nonacute complications associated with interscalene block and shoulder surgery: a prospective study. Anesthesiology. 2001 Oct;95(4):875-80. doi: 10.1097/00000542-200110000-00015. PMID 11605927
- [Background] Fredrickson MJ, Kilfoyle DH. Neurological complication analysis of 1000 ultrasound guided peripheral nerve blocks for elective orthopaedic surgery: a prospective study. Anaesthesia. 2009 Aug;64(8):836-44. doi: 10.1111/j.1365-2044.2009.05938.x. PMID 19604186
- [Background] Jeng CL, Torrillo TM, Rosenblatt MA. Complications of peripheral nerve blocks. Br J Anaesth. 2010 Dec;105 Suppl 1:i97-107. doi: 10.1093/bja/aeq273. PMID 21148659

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL 1.3 % in 20 ML Injection: EXPAREL (bupivacaine liposome injectable suspension, 20 mL single use vial, 1.3% [13.3 mg/mL]) is a liposome injection of bupivacaine, an amide local anesthetic, indicated for single-dose infiltration into the surgical site to produce postsurgical analgesia. EXPAREL dosage is based on the following factors:
  * size of surgical site
  * volume required to cover the area
  * individual patient factors that may impact the safety of an amide local anesthetic
  * maximum doe of 266 mg (20 mL)
  EXPAREL 1.3 % in 20 ML Injection: EXPAREL single shot dose given as an analgesia for arthroscopic rotator cuff repair surgery.
Period: Overall Study
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
Number analyzed (Participants) | 13
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 56.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: VAS Pain Score
Description: Patient reported numeric pain rating using visual analog scale (VAS) (0 = none, 10 = severe)
Time Frame: 12 hours, 24 hours, 36 hours, 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
Number analyzed (Participants) | 13
units on a scale
  12 Hours | 2.7 (3.0)
  24 Hours | 3.2 (3.5)
  36 Hours | 2.3 (2.7)
  48 Hours | 2.1 (2.6)

2. Primary Outcome: Narcotic Medication Usage
Description: Number of narcotic medication tablets consumed
Time Frame: 12 hours, 24 hours, 36 hours, 48 hours, 3 days, 7 days, 14 days
Measure: Mean (Standard Deviation); unit: quantity of tablets
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
Number analyzed (Participants) | 13
quantity of tablets
  12 Hours | 1.38 (1.67)
  24 Hours | 1.54 (2.06)
  36 Hours | 1.68 (2.08)
  48 Hours | 1.36 (1.44)
  Day 3 | 8.18 (9.75)
  Day 7 | 14.42 (16.45)
  Day 14 | 18.02 (20.07)

3. Secondary Outcome: American Shoulder and Elbow Surgeons Shoulder Score (ASES) on Surgical Arm
Description: American Shoulder and Elbow Surgeons Shoulder Score (ASES) of surgical arm measured utilizing patient reported outcome surveys. (0 = no function; 100 = full function)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
Number analyzed (Participants) | 13
score on a scale | 48.8 (7)

4. Secondary Outcome: American Shoulder and Elbow Surgeons Shoulder Score (ASES) of Healthy Arm
Description: American Shoulder and Elbow Surgeons Shoulder Score (ASES) of healthy (nonsurgical) arm measured utilizing patient reported outcome surveys. (0 = no function; 100 = full function)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Arm: Measurement of healthy arm against that of the surgical arm which received the EXPAREL injection.
Arm/Group | Healthy Arm
Number analyzed (Participants) | 13
score on a scale | 73.6 (23.7)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | EXPAREL 1.3 % in 20 ML Injection
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No